CLINICAL TRIAL: NCT00418067
Title: Comparison of the Efficacy and the Safety of Zotarolimus-Eluting Stent Versus Sirolimus-Eluting Stent and PacliTaxel-Eluting Stent for Coronary Lesions
Brief Title: Zotarolimus-Eluting Stent Versus Sirolimus-Eluting Stent and PacliTaxel-Eluting Stent for Coronary Lesions
Acronym: ZEST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seung-Jung Park (Other)
Collaborators: Medtronic Vascular (Industry)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, Comparison of the Efficacy of Zotarolimus(ABT 578)-Eluting Stent versus Sirolimus-Eluting Stent versus Paclitaxel-Eluting Stent for Coronary Lesions: The Prospective, Randomized, and Multi-center Trial, CardioVascular Research Foundation, Korea
Organization: CardioVascular Research Foundation, Korea (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2006-0136
Record Dates: First submitted 2007-01-03; First posted 2007-01-04 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2012-08

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Stent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cypher (Active Comparator): Sirolimus-eluting stent
  Interventions: Device: Cypher
- Taxus Liberte (Active Comparator): Paclitaxel-eluting stent
  Interventions: Device: Taxus Liberte
- Endeavor (Experimental): Zotarolimus-eluting stent
  Interventions: Device: Endeavor

INTERVENTIONS:
Device: Endeavor — Zotarolimus-eluting stent
  Other Names: Zotarolimus-eluting stent
  Arms: Endeavor
Device: Cypher — Sirolimus-eluting stent
  Other Names: Sirolimus-eluting stent
  Arms: Cypher
Device: Taxus Liberte — Paclitaxel-eluting stent
  Other Names: Paclitaxel-eluting stent
  Arms: Taxus Liberte

SUMMARY:
The purpose of this study is to establish the safety and long-term effectiveness of coronary stenting with the ABT 578-eluting balloon expandable stent (Medtronic, Minneapolis, MN) vs. the sirolimus-eluting balloon expandable stent (Cordis Johnson & Johnson, Warren, New Jersey) and the paclitaxel-eluting stent (Taxus liberte, Boston Scientific) for the treatment of coronary stenosis in routine clinical practice.

DETAILED DESCRIPTION:
Previous studies have documented that a slow-release polymeric sirolimus-eluting stent (Cypher, Cordis) and paclitaxel-eluting stent (Taxus, Boston Scientific) reduce neointimal formation and result in decrease of angiographic restenosis and target lesion revascularization at 1-3 years in the multicenter randomized clinical trials RAVEL, SIRIUS, and TAXUS I-VI.From these studies, the two leading drug-eluting stents (DESs) of the Cypher and Taxus have been widely and rapidly accepted as a standard treatment of coronary lesions.

Recently, randomized studies were conducted to reveal different outcomes of the different two DESs. These studies showed that the sirolimus-eluting stent was better than the paclitaxel-eluting stent in terms of lower angiographic restenosis rate or the two DESs were similar in angiographic outcomes. A recent meta-analysis supported results of the former randomized studies. Patients receiving sirolimus-eluting stent had a significantly lower risk of restenosis and target vessel revascularization compared with those receiving paclitaxel-eluting stent.

With a recent approval of new DES, ABT-578-eluting stent (Endeavor, Medtronic, Minneapolis, MN), other comparison studies have been conducted to compare Endeavor ABT-578-eluting stent with the sirolimus-eluting stent and paclitaxel-eluting stent. ABT-578 and sirolimus share some common structural and biological properties. The ENDEAVOR clinical trials are currently in progress to evaluate a phosphoryl choline (PC)-coated ABT-578-eluting stent for the prevention of restenosis. The Endeavor ABT-578-eluting stent utilizes a cobalt alloy balloon-expandable stent (Driver; Medtronic) with a geometry similar to the stainless steel stent used in this preliminary study (S7; Medtronic). The Endeavor ABT-578-eluting stent also employees a PC strut surface coating as the drug delivery reservoir with a dose of 10 ug/mm of ABT-578. The Endeavor ABT-578-eluting stent, however, differs from the stent used in this experimental study by the addition of a drug-free PC coating to serve as a diffusion barrier to retard drug release from the polymer reservoir. Angiographic analysis at 4 months in the 100-patient focal de novo lesion ENDEAVOR I feasibility study demonstrated a mean in-stent percent diameter stenosis of approximately 14% and a late lumen loss of 0.3 mm with a low frequency of target lesion revascularization (1%). The clinical outcomes from the ENDEAVOR II (1,500 patients randomized to ABT-578 or bare metal stent) and the ENDEAVOR III (436 patients randomized 3:1 to ABT-578 or Cypher) trials as well as other ongoing studies showed efficacy of the PC-coated ABT-578-eluting stent. In ENDEAVOR III study, the Endeavor stent had larger late loss and higher binary restenosis in both the analysis segment and stented segment. In contrast, the TLR rates are not statistically different between the Endeavor (6.0%) and the Cypher (5.3%, p=1.0) stents. This result of this study raised several questions to warrant further randomized studies 1) is the angiographic superiority of Cypher stent applied to the more complex lesions, 2) why is the TLR rate similar in spite of significantly different angiographic outcomes, 3) which is better in the Endeavor and the Taxus stents, etc. The ENDEAVOR IV study is being conducted to compare the safety and efficacy of the Endeavor stent versus the Taxus stent. However, the inclusion of ENDEAVOR IV study was also limited that this study did not include all complex lesions. Because of the limitations of current ENDEAVOR series, a further large randomized study for the concurrent comparison of the three DESs in the treatment of real-world practice would be needed.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be at least 18 years of age.
* Significant coronary artery stenosis (>50% by visual estimate)
* Patients with stable (CCS class 1 to 4) or acute coronary syndromes (unstable angina pectoris class IB, IC, IIB, IIC, IIIB, IIIC or NSTEMI) or patients with atypical chest pain or without symptoms but having documented myocardial ischemia, amenable to stent-assisted percutaneous coronary intervention
* The patient or guardian agrees to the study protocol and the schedule of clinical and angiographic follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site.

Exclusion Criteria:

* The patient has a known hypersensitivity or contraindication to any of the following medications:

  • Heparin, Aspirin, Both Clopidogrel and Ticlopidine, Sirolimus, paclitaxel, ABT 578, Stainless steel and/or Contrast media (patients with documented sensitivity to contrast which can be effectively pre-medicated with steroids and diphenhydramine [e.g. rash] may be enrolled. Patients with true anaphylaxis to prior contrast media, however, should not be enrolled).
* Female of childbearing potential, unless a recent pregnancy test is negative, who possibly plan to become pregnant any time after enrollment into this study.
* Current known current platelet count <100,000 cells/mm3 or Hgb <10 g/dL.
* An elective surgical procedure is planned that would necessitate interruption of antiplatelet drugs during the first 12 months post enrollment.
* Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment).
* Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period.
* Patients who have target lesion of in-stent restenosis at the stented segment of drug-eluting stent (in-stent restenosis of bare metal stent can be included).
* Patients with EF<30%.
* Patients with cardiogenic shock
* Acute STEMI patients within symptom onset < 12 hours needing primary angioplasty
* Creatinine level > 3.0mg/dL or dependence on dialysis.
* Severe hepatic dysfunction (AST and ALT > 3 times upper normal reference values).
* Patients with left main stem stenosis (>50% by visual estimate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2645 (Actual)
Dates: Start 2006-10; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
The composite of death (all cause-mortality), myocardial infarction, and ischemia-driven target vessel revascularization | at 12 months after the index procedure

SECONDARY OUTCOMES:
All-cause Death | In-hospital, 30 days, 6 months, 1 year, and thereafter annually upto 5 years
Cardiac death | In-hospital, 30 days, 6 months, 1 year, and thereafter annually upto 5 years
Myocardial infarction | In-hospital, 30 days, 6 months, 1 year, and thereafter annually upto 5 years
Target vessel revascularization (all and ischemia-driven) | In-hospital, 30 days, 6 months, 1 year, and thereafter annually upto 5 years
Target lesion revascularization (all and ischemia-driven) | In-hospital, 30 days, 6 months, 1 year, and thereafter annually upto 5 years
Stent thrombosis by definition of Academic Research Consortium (ARC) | In-hospital, 30 days, 6 months, 1 year, and thereafter annually upto 5 years
Late luminal loss in both in-stent and in-segment | at 8 month angiographic follow-up
Binary restenosis in both in-stent and in-segment | At 8 month angiographic follow-up
Procedural success defined as achievement of a final diameter stenosis of <30% by QCA using any percutaneous method, without the occurrence of death, Q wave MI, or urgent revascularization during the hospital stay. | In-hospital

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jung Park, MD, PhD, Principal Investigator — Department of Medicine, Asan Medical Center, University of Ulsan College of Medicine
Locations (20):
- South Korea (20):
  - Soonchunhyang University Bucheon Hospital, Bucheon-si
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook National University Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - Asan Medical Center, Gangneung
  - Chonnam National University Hospital, Gwangju
  - NHIC Ilsan Hospital, Ilsan
  - Chonbuk National University Hospital, Jeonju
  - Pusan Natioanal University Hospital, Pusan
  - Hallym University Sacred Heart Hospital, Pyeongchon
  - Seoul National University Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Korea University Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - St.Mary's Catholic Medical Center, Seoul
  - Yonsei University Medical Center, Seoul
  - Ajou University Hospital, Suwon
  - Ulsan University Hospital, Ulsan
  - Yonsei University Wonju Christian Hospital, Wŏnju

REFERENCES:
- [Derived] Kang SJ, Mintz GS, Park DW, Lee SW, Kim YH, Lee CW, Han KH, Kim JJ, Park SW, Park SJ. Comparison of zotarolimus-eluting stents with sirolimus-eluting and paclitaxel-eluting stents: intimal hyperplasia and vascular changes assessed by volumetric intravascular ultrasound analysis. Circ Cardiovasc Interv. 2011 Apr 1;4(2):139-45. doi: 10.1161/CIRCINTERVENTIONS.110.957936. Epub 2011 Mar 1. PMID 21364151
- [Derived] Park DW, Kim YH, Yun SC, Kang SJ, Lee SW, Lee CW, Park SW, Seong IW, Lee JH, Tahk SJ, Jeong MH, Jang Y, Cheong SS, Yang JY, Lim DS, Seung KB, Chae JK, Hur SH, Lee SG, Yoon J, Lee NH, Choi YJ, Kim HS, Kim KS, Kim HS, Hong TJ, Park HS, Park SJ. Comparison of zotarolimus-eluting stents with sirolimus- and paclitaxel-eluting stents for coronary revascularization: the ZEST (comparison of the efficacy and safety of zotarolimus-eluting stent with sirolimus-eluting and paclitaxel-eluting stent for coronary lesions) randomized trial. J Am Coll Cardiol. 2010 Oct 5;56(15):1187-95. doi: 10.1016/j.jacc.2010.03.086. PMID 20883925